CLINICAL TRIAL: NCT01858194
Title: REnal Sympathetic dEnervaTion as an a Adjunct to Catheter-based VT Ablation
Acronym: RESET-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 13-1462
Record Dates: First submitted 2013-03-19; First posted 2013-05-21 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Ventricular Tachycardia
Keywords: Tachycardia, Renal Sympathetic Denervation; Catheter Ablation; Cardioverter-Defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal sympathetic denervation (Experimental): Catheter-based Renal Sympathetic Denervation Ablation Arm
  Interventions: Device: Renal sympathetic denervation
- VT ablation alone (Placebo Comparator): No further therapy in addition to VT ablation
  Interventions: Device: VT ablation alone

INTERVENTIONS:
Device: Renal sympathetic denervation — * The ablation catheter is placed within a long vascular sheath and advanced into the renal artery. The sheath is advanced over the catheter to engage the renal artery ostium and allow for contrast injection and visualization of the vessel during catheter manipulation.
  * After completion of the measurement, no more than six radiofrequency ablation lesions separated both longitudinally and rotationally (a "spiral pattern", see figure) will be placed per renal artery. The power will be started at 10 W and titrated to a maximum 20 W, as deemed appropriate by the impedance drop (goal 10% drop). Each lesion should be between 30-120 seconds in duration (no more than 120 seconds per lesion).
  Other Names: Ablation Arm; Catheter-based Renal Sympathetic Denervation
  Arms: Renal sympathetic denervation
Device: VT ablation alone — Placebo arm will receive standard VT ablation using current techniques
  Arms: VT ablation alone

SUMMARY:
Despite significant advances in the management of ventricular arrhythmias through the use of ICD therapy, AADs, and catheter-based ablation strategies, considerable challenges remain. The optimal method for the prevention of recurrent VT following catheter ablation remains unclear. RSDN may be an effective tool for preventing ventricular arrhythmias, and associated ICD therapies, by reducing central sympathetic tone, catecholamine levels, and the renin-angiotensin- aldosterone system and promoting ventricular remodeling. Although RSDN has been shown to reduce the recurrence of VT in a case report of 2 patients suffering from electrical storm, to date no large prospective randomized study has evaluated the impact of RSDN in the prevention of recurrent VT in patients following catheter ablation of VT with ischemic or non-ischemic ventricular dysfunction. This study will specifically evaluate the safety and efficacy of adjunctive RSDN in the prevention of ICD therapy in patients with ischemic or non-ischemic ventricular dysfunction who are to receive a catheter-based VT ablation.

DETAILED DESCRIPTION:
The goal of this trial is to test the impact of catheter-based renal sympathetic denervation (RSDN) as an adjunctive treatment for patients with either ischemic or non-ischemic cardiomyopathy undergoing catheter ablation of ventricular tachycardia (VT). The proposed study is a prospective, multicenter, randomized control trial. Patients undergoing VT ablation will be randomized to either VT ablation alone or VT ablation + RSDN.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Structural heart disease (post-MI, dilated cardiomyopathy, sarcoid myopathy, hypertrophic cardiomyopathy, chagas-related cardiomyopathy, etc.)
* Planned for catheter-based ablation of VT
* All patients will have an existing ICD
* Accessibility of renal vasculature (determined by renal angiography)
* Ability to understand the requirements of the study
* Willingness to adhere to study restrictions and comply with all post- procedural follow-up requirements

Exclusion Criteria:

* MI or CVA within 30 days
* Coronary Artery Bypass Graft (CABG) within 30 days of this procedure
* Known renovascular abnormalities that would preclude RSDN (eg, renal artery stenosis)
* GFR <30 ml/min (unless receiving dialysis)
* Life expectancy <1 year for any medical condition
* Any condition resulting in a contraindication to anticoagulation (e.g. GI bleeding)
* Inability to give informed consent
* Known pregnancy or positive -HCG within 7 days of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Y Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Homolka Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 participants received ID numbers because they were consented. 3 patients were screen failures due to accessibility of renal vasculature and Investigator discretion.
  1 patient was a non-randomized roll- in where data was not collected.
Groups:
- Renal Sympathetic Denervation: Catheter-based Renal Sympathetic Denervation Ablation Arm
  Renal sympathetic denervation: • The ablation catheter is placed within a long vascular sheath and advanced into the renal artery. The sheath is advanced over the catheter to engage the renal artery ostium and allow for contrast injection and visualization of the vessel during catheter manipulation.
  • After completion of the measurement, no more than six radiofrequency ablation lesions separated both longitudinally and rotationally (a "spiral pattern", see figure) will be placed per renal artery. The power will be started at 10 W and titrated to a maximum 20 W, as deemed appropriate by the impedance drop (goal 10% drop). Each lesion should be between 30-120 seconds in duration (no more than 120 seconds per lesion).
Period: Overall Study
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Started | 8 | 9
Completed | 8 (All patients in Control arm completed.) | 7
Not Completed | 0 | 2
Not completed — Total Artificial Heart Implant | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.73) | 56.78 (9.43) | 58.88 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 3 | 7 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Freedom From First Event Requiring ICD Therapy
Description: Probability of freedom from first event requiring ICD therapy at 12 months and at 24 months
Time Frame: 24 months
Measure: Number; unit: probability of freedom
Arm/Group | Renal Sympathetic Denervation | VT Ablation Alone
Number analyzed (Participants) | 9 | 8
probability of freedom
  12 months | 62.5 | 50
  24 months | 62.5 | 37.5

2. Secondary Outcome: Number of Appropriate ICD Shocks for Ventricular Arrhythmia
Description: An Appropriate ICD therapy is defined as anti-tachycardia pacing (ATP) or shock therapy for ventricular tachycardia or fibrillation.
Time Frame: at 24 months
Measure: Number; unit: occurrences
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
occurrences | 7 | 12

3. Secondary Outcome: Number of Inappropriate ICD Therapy
Description: Number of inappropriate ICD therapy including both appropriate and inappropriate shocks
Time Frame: at 24 months
Measure: Number; unit: occurrences
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
occurrences | 5 | 7

4. Secondary Outcome: All ICD Therapies (Appropriate + Inappropriate)
Description: cumulative ICD therapies including both appropriate and inappropriate shocks
Time Frame: 24 months
Measure: Number; unit: occurrences
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
occurrences | 32 | 32

5. Secondary Outcome: Number of Participants With Mortality, ICD Storm and Incessant VT
Description: Number of Participants with a composite of Mortality, ICD storm, and Incessant VT
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
Participants | 1 | 3

6. Secondary Outcome: Number of Participants With Hospitalizations for Cardiovascular Causes
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
Participants | 3 | 1

7. Secondary Outcome: Number of Episodes of Total VT Burden
Description: Total VT burden (Number of episodes)
Time Frame: at 24 months
Measure: Number; unit: episodes
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
episodes | 20 | 12

8. Secondary Outcome: Number of Participants With All-Cause Mortality
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Occurrences of ICD Storm
Description: The occurrence of ICD storm, defined as ≥3 appropriate shock therapies within 24 hours.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
Participants | 1 | 3

10. Secondary Outcome: Change in Brain Natriuretic Peptide (BNP)
Description: Differences in blood hormone measurements as measured by BNP as compared on 12 months to baseline.
Time Frame: at baseline and at 12 months
Population: results only for those participants who have both timepoint data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 3 | 2
mg/dL | -12.33 (46.6) | -2.5 (24.75)

11. Secondary Outcome: Differences in BUN/Creatinine Measurements
Description: Differences in BUN/creatinine measurements compared at 12 months to baseline.
Time Frame: baseline and 12 months
Population: Results only available for participants with data for both timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 4 | 3
mg/dL
  BUN | -4 (4.84) | 1.67 (5.68)
  Creatinine | 0.095 (0.24) | .04 (.03)

12. Secondary Outcome: Change in LV Size
Description: LV size measured by trans-thoracic echocardiography, as compared at 12 months to baseline
Time Frame: baseline and 12 months
Population: Results only available for participants with data for both timepoints.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 4 | 1
cm | -.125 (.59) | -1.4 (NA) — data for N=1

13. Secondary Outcome: Number of Procedure-related Adverse Events
Description: Procedure related adverse events including, but not limited to hematomas, pseudoaneurysms, renal artery stenosis, renal impairment, thromboembolic events, stroke, pericardial bleeding including tamponade and myocardial infarction.
Time Frame: 24 months
Measure: Number; unit: events
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
events | 3 | 3

14. Secondary Outcome: Changes in Mean Arterial Pressure
Description: Change in mean arterial pressure
Time Frame: baseline and 24 months
Population: Results only available for participants with data for both timepoints.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 6 | 5
mmHg | 3.33 (8.41) | 13.77 (18.75)

15. Secondary Outcome: Number of Participants With Orthostatic Hypertension
Description: Number of participants with other individual complication rates specifically orthostatic hypertension
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Other Complications
Description: Other individual complication rates including, but not limited to MI and death
Time Frame: at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
Participants | 1 | 2

17. Secondary Outcome: Number of Occurrences of Major Complication Rate
Description: 30-day Major Complication Rate defined as death, stroke, MI or any other serious adverse events related to the treatment or procedure within the first 30 days or through hospital discharge (whichever is longer)
Time Frame: 30 days
Measure: Number; unit: occurrences
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 8 | 9
occurrences | 2 | 3

18. Secondary Outcome: Procedure Time
Description: Renal Denervation Procedure time
Time Frame: during procedure
Population: Results only for those participants who underwent renal sympathetic denervation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | VT Ablation Alone | Renal Sympathetic Denervation
Number analyzed (Participants) | 0 | 9
minutes |  | 27.83 (8.8)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Renal Sympathetic Denervation | VT Ablation Alone
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/8
Other Adverse Events (participants affected / at risk) | 5/9 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Sympathetic Denervation (N=9) | VT Ablation Alone (N=8)
VT recurrence (Cardiac disorders) | 0 | 2
Non-sustained VT (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Macrohematuria (Renal and urinary disorders) | 0 | 1
AF with urosepsis (General disorders) | 1 | 0
Worsening heart failure/Total artifical heart implant (Cardiac disorders) | 1 | 0
Pseudoaneurysm at septal aspect of LV apex (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Sympathetic Denervation (N=9) | VT Ablation Alone (N=8)
VT recurrence (Cardiac disorders) | 0 | 2
Dissection of left external iliac artery (Cardiac disorders) | 0 | 1
Paresthesia (Skin and subcutaneous tissue disorders) | 0 | 1
LUE Cephalic vein thrombosis (Vascular disorders) | 1 | 0
Hypotension with pleuritic chest pain (Cardiac disorders) | 1 | 0
Kidney pain with near syncope (Hepatobiliary disorders) | 1 | 0
Flu (Infections and infestations) | 1 | 0
Bradycardia associated with dyspnea on exertion (Cardiac disorders) | 1 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT01858194/Prot_SAP_000.pdf